CLINICAL TRIAL: NCT04843150
Title: Pharmacokinetics and Immunogenicity of the First Doses of PEG-Asparaginase -An ALLTogether Pilot Study
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Klug Albertsen, M.D., PhD, Associate Professor, Aarhus University Hospital
Other Study IDs: A2G-pilot-asp
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common malignant disease in childhood. Survival rates exceed 90% in children and 75% in adults (aged 18-45 years). During the induction period Asparaginase is an indispensable part of the multiagent treatment, but is often associated with hypersensitivity, either with clinical allergy or silent inactivation. In both cases, Asparaginase is inactivated. It is well known that truncation of Asparaginase treatment due to inactivation reduces survival. To approach understanding Asparaginase dynamics and hypersensitivity in ALL patients it is important to examine the pharmacokinetics of Asparaginase.

The aim of this study is to identify serological parameters for prediction of hypersensitivity reaction after the first doses of PEG-Asparaginase given intravenously on the ALLTogether protocol.

DETAILED DESCRIPTION:
Asp enzyme activity is measurable in plasma, and trough levels above 100 IU/l secure effect. Patients, who have their treatment truncated, have inferior outcome. For many years prolonged Asp treatment for 30 weeks has been part of most protocols worldwide, but a recent Nordic randomized study showed that less asparaginase (8 doses vs 15 doses intramuscularly (IM)) results in the same disease-free survival and significant less toxicity in the less intensive treatment arm (6).

Accordingly, in the current Western European protocol (ALLTogether) less Asp is now given. The Nordic Countries participate in this protocol.

Unlike in the previous Nordic protocol, NOPHO ALL2008, in ALLTogether Asp will be initiated early during induction (day 4 compared to day 30) and given intravenously (IV) and not IM. In February 2017 it was approved by the NOPHO Board to do more extensive pharmacokinetic studies of IM administered PEG-asparaginase, as it has not been shown if IM or IV is preferably in respect to minimizing the incidence of hypersensitivity. Most study groups in the world use IV administration, thus NOPHO has a unique chance to illuminate inactivation after IM administration, also in adult patients. Other groups have not published this.

For >50% of the patients in ALLTogether, the induction therapy has been reduced from 4 drugs to 3 drugs. This emphasizes the importance of optimal treatment from the beginning. Therapeutic Drug Monitoring (TDM) will identify patients without activity in order to change Asp preparation. Additional sampling close after the first dose of PEG-Asp is expected to identify these patients earlier, providing an opportunity to optimize their treatment for better disease-free survival.

The aim of this study is to identify serological parameters for prediction of hypersensitivity reaction after the first dose of PEG-Asp given IV on the ALLTogether protocol.

ELIGIBILITY:
Inclusion Criteria:

* Treated for acute lymphoblastic leukemia (ALL) on the ALL2GETHER pilot protocol

Exclusion Criteria:

* none

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients with ALL 1-45 years of age treated on the ALLTOGETHER pilot protocol in the Nordic and Baltic countries.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with hypersensitivity Clinical allergy / silent inactivation | 2018-2021
  Patients with allergic reactions or silent inactivation

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte K Albertsen, MD, Principal Investigator — M.D., PhD, Associate Professor, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Pediatrics, Skejby Hospital, Aarhus
  - Aarhus University Hospital, Denmark, Aarhus N

IPD SHARING:
Plan to Share IPD: Undecided